CLINICAL TRIAL: NCT06947018
Title: Impact Evaluation of Türkiye's Adolescent Girls' and Boys' Empowerment Programme for Elimination of Child Marriage
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNICEF (Other)
Responsible Party: Principal Investigator, Yasemin Kisbu, Impact Evaluation Consultant, UNICEF
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HML2855
Record Dates: First submitted 2025-04-07; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Marriage Age; Marriage
Keywords: Child marriage; Adolescent empowerment; Refugees; Life skills

STUDY DESIGN:
Intervention Model Description: The trial is an individually randomized intervention study where the intervention versus a control group is allocated on a 1:1 basis to households (adolescent girls, boys and their caregivers), stratified by study site (Istanbul, Ankara, Izmir, Adana, Gaziantep, and Hatay) and nationality (Syrian refugees versus Turkish nationals). The intervention group receives the Adolescent Girls' and Boys' Empowerment for Elimination of Child Marriage intervention, whereas the control group is a delayed treatment group who will be offered the intervention upon completion of the trial and follow-up data collection (if funding allows).
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be masked at baseline only, as there is no placebo treatment, thus participants will know their status by follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adolescent Girls' and Boys' Empowerment Program (Experimental): Adolescent Girls' and Boys' Empowerment Program for Elimination of Child Marriage
  Interventions: Behavioral: Adolescent Girls' and Boys' Empowerment Program
- Control (No Intervention): Business as usual (delayed intervention, post-trial - if funding allows)

INTERVENTIONS:
Behavioral: Adolescent Girls' and Boys' Empowerment Program — The program was developed based on a social behavioural change (SBC) approach in order to change attitudes and behaviours of the participants, consisting of the following main activities on a 6 - 8 week cycle.
  * Girls' Empowerment Training: Workshops comprise six sessions of approximately 80 minutes each, held separately with girls aged 12-15 and 16-18 years in groups of approximately 12-20 adolescents on a range of life skill themes.
  * Boys' Awareness Raising Training: Similar to the girls' training, four workshops are organized for boys aged 12-15 and 16-18 years, in separate sessions, with similar length and group size.
  * Awareness Raising Seminars to Caregivers: Caregivers (e.g., mothers, fathers) are invited to a one-time seminar focused on the negative outcomes of child marriage and role of caregivers in preventing child marriage, lasting approximately one hour and conducted separately for fathers and mothers to eventually influence social norms in the family and communities.
  Arms: Adolescent Girls' and Boys' Empowerment Program

SUMMARY:
Low income, refugee, displaced and disaster affected populations face a variety of protection risks, including higher risk of child, early and forced marriage and unions (CEFMU). This is the case in Türkiye, where low income, refugee populations and those affected by the 2023 earthquake in Southern and Central Türkiye face elevated risk of child marriage. As part of the UNICEF Türkiye Country Office (TCO) commitment to implement comprehensive interventions that aim to contribute to a change in social norms and attitudes towards gender equality, the CO and partners have developed the "Adolescent Girls' and Boys' Empowerment for Elimination of Child Marriage" program (hereafter "the program"). The program is an 8-week group-based empowerment and life skills training for adolescent girls aged 12 - 18 years old, a 4-session adolescent boys awareness training, and a one-time awareness raising seminar for caregivers. The current trial has the overall objective of evaluating the short-term causal impact of the program with respect to CEFMU and related outcomes for adolescent girls. The trial design is an individual randomized control trial, allocating 820 households with adolescent girls to either treatment or control on a 1:1 basis. The primary data collection includes a pre- and post-intervention caregiver and adolescent face-to-face survey, as well as a one-time qualitative data collection. The trial results will inform the future operation and scale-up of the program, as well as contribute to the broader evidence base on what works to increase the empowerment of adolescent girls and reduce CEFMU.

DETAILED DESCRIPTION:
Low income, refugee, displaced and disaster affected populations face a variety of protection risks, including higher risk of child, early and forced marriage and unions (CEFMU). This is the case in Türkiye, where low income, refugee populations and those affected by the 2023 earthquake in Southern and Central Türkiye face elevated risk of child marriage. As part of the UNICEF Türkiye Country Office (TCO) commitment to implement comprehensive interventions that aim to contribute to a change in social norms and attitudes towards gender equality, the CO and partners have developed the "Adolescent Girls' and Boys' Empowerment for Elimination of Child Marriage" program (hereafter "the program"). The program is an 8-week group-based empowerment and life skills training for adolescent girls aged 12 - 18 years old, a 4-session adolescent boys awareness training and a one-time awareness raising seminar for caregivers. The current trial has the overall objective of evaluating the short-term causal impact of the program with respect to CEFMU and related outcomes for adolescent girls. The trial seeks to answer the following evaluation questions:

* 1) Does the program improve participant adolescent girls' agency, self-confidence, and gender-equitable attitudes (including for CEFMU), and to what extent?
* 2) Does the program improve the household enabling environment, including gender-equitable attitudes (including CEFMU), social support, protective behaviors against CEFMU, and use of social services among participating caregivers and in the broader community, and to what extent?
* 3) Does the program reduce CEFMU for adolescent girls, and to what extent?
* 4) Through which pathways (or combination of pathways) do potential impacts occur?
* 5) Was the program implemented in a manner to maximize potential impacts? and
* 6) What is the return-on-investment (cost-benefit calculation) for the program? The trial design is an individual randomized control trial, allocating 820 households with adolescent girls to either treatment or control on a 1:1 basis. The primary data collection includes a pre- and post-intervention caregiver and adolescent face-to-face survey, as well as a one-time qualitative data collection. The trial results will inform the future operation and scale-up of the program, as well as contribute to the broader evidence base on what works to increase the empowerment of adolescent girls and reduce CEFMU.

ELIGIBILITY:
Inclusion criteria (primary study participant, however note that primary female caregivers and siblings will be invited to participate in the study pending inclusion of primary study participant):

* Adolescent girls aged 12 - 17 years
* Unmarried girls
* Have never previously been exposed to the intervention
* Live in a family or household with at least one adult caregiver
* Live in a family who are social service clients of the implementing partner
* Live in a family who are risk-assessed as 'low' or 'medium' on the family risk assessment tool
* Live in a family which is planning on staying in the catchment area of the intervention in the subsequent 6-months

Exclusion criteria:

* Adolescent girls younger than 12 or older than 17 years
* Girls who are married or cohabiting
* Previously been exposed to the intervention
* Are in institutionalized or non-family-based care
* Live in a family who are not social service clients of the implementing partner
* Live in a family who are risk-assessed as 'high' or 'highest' on the family risk assessment tool
* Live in a family which is planning on moving outside the catchment area of the intervention in the subsequent 6-months

Ages: 12 Years to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 820 (Estimated)
Dates: Start 2025-04-21 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of girls married or cohabiting | Baseline and 8-weeks post-intervention
  Marriage or cohabitation status measured among adolescent girls
Score on new general self-efficacy scale (short form, higher is better) | Baseline and 8-weeks post-intervention
  Eight-item scale asking about internal efficacy, with response options on a five-point scale, ranging from 1 = strongly disagree, to 5 = strongly agree (score ranges from 8 - 40). Widely used scale for individual ability to achieve goals across a range of different situations, despite difficulties. Interpreted as a sub-component of the construct of adolescent girls' agency.
Score on decision-making scale (higher is better) | Baseline and 8-weeks post-intervention
  Ten-item scale asking about freedom to make choices across domains, with response options on a four-point scale, ranging from 1 = not at all, to 4 = a large extent (score ranges from 10 - 40). Adapted from the program version of the women's empowerment in agriculture index (pro-WEAI) to include adolescent-specific questions, previously piloted in Ethiopia among male and female youth. Interpreted as a sub-component of the construct of adolescent girls' agency.
Score on voice scale (higher is better) | Baseline and 8-weeks post-intervention
  Eight-item scale asking about girls' ability to share feelings and speak up in different scenarios, with response options on a four-point scale, ranging from 1 = never, to 4 = all of the time (score ranges from 8 - 32). Voice scale is adapted from Global Early Adolescent Survey and interpreted as a sub-component of the construct of adolescent girls' agency.
Score on child marriage attitudes scale (higher is better) | Baseline and 8-weeks post-intervention
  Thirteen-item scale developed and piloted in Türkiye by the author team to measure child marriage attitudes, with response options on a four-point scale, ranging from 1 = strongly disagree to 4 = strongly agree. The scale is measured among adolescent girls and boys, as well as their caregivers (score ranges from 13 - 52).

SECONDARY OUTCOMES:
Scale of perceived social support (higher is better). | Baseline and 8-weeks post-intervention
  The family and friends' sub-scales of the multi-dimensional scale of perceived social support (MSPSS) consisting of nine questions answered on a four-point scale, ranging from 1 = strongly disagree to 4 = strongly agree. The scale is measured among adolescent girls and ranges from 9 - 36.
The Balanced Cohesion subscale of the Family Adaptability and Cohesion Evaluation Scale (higher is better) | Baseline and 8-weeks post-intervention
  The Balanced Cohesion subscale of the Family Adaptability and Cohesion Evaluation Scale is a seven-item scale answered on a five-point scale, ranging from 1 = strongly disagree to 5 = strongly agree. The scale is measured among caregivers and ranges from 7 - 35.
The Revised Family Communication Pattern Instrument Conversation Orientation Sub-scale (higher is better) | Baseline and 8-weeks post-intervention
  The Revised Family Communication Pattern Instrument Conversation Orientation Sub-scale measures parent-adolescent communication and is a 15-item scale answered on a five-point scale, ranging from 1 = strongly disagree to 5 = strongly agree. The scale is administered to caregivers and ranges from 15 - 75.
Score on willingness to intervene and speak out for girls' scale (higher is better) | Baseline and 8-weeks post-intervention
  Willingness to speak out and take action to support girls measured using simple self-reported questions on willingness to speak up against harmful behaviors: 1) child marriage, 2) violence against girls, 3) girls' rights and 4) for girls in times of need. These four domains are each assessed using one question answered on a four-point scale, ranging from 1 = strongly disagree to 4 = strongly agree. The scale is measured among adolescent boys and caregivers and ranges from 4 - 32.
Linkages to services scale (higher is better) | 8-weeks post-intervention
  Received assistance or benefits from services measured among adolescent girls and caregivers, collected as a simple sum = 1 if received any services from: 1) health, 2) social, or 3) legal services (ranges from 0 - 3)

CONTACTS AND LOCATIONS:
Overall Officials: Zlata Bruckauf, Ph.D., Study Director — UNICEF
Locations (1):
- UNICEF Türkiye, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data from the trial will be owned by UNICEF and efforts will be made to share the deindentified data in a public repository, pending UNICEF approval. In addition, it is expected that de-identified replication files will be made publicly available upon the publication of any journal articles to allow the reproduction of all tables, figures and results, alongside statistical replication code.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: IPD will be available 24 months after the trial ends, or upon publication of the main trial results, with no end date projected.
Access Criteria: It is expected that data will be accessible to all the scientific community via open repository.